CLINICAL TRIAL: NCT06930716
Title: Use of Paired Vagus Nerve Stimulation in Mobilization of Patients With Prolonged Disorders of Consciousness: A Pilot Feasibility Study
Brief Title: Paired Vagus Nerve Stimulation in Mobilization of Patients With Prolonged Disorders of Consciousness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jenna Mancuso, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-01339
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-04

CONDITIONS: Consciousness Disorders; Brain Injury; Altered Level of Consciousness
Keywords: Therapy; Rehabilitation; Neuromodulation
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with Prolonged Disorders of Consciousness (pDOC) (Experimental): Patients with pDOC receiving paired transauricular vagus nerve stimulation (taVNS) and robotic tilt table mobilization (RTTM) to maximize functional recovery,
  Interventions: Device: Transcutaneous vagus nerve stimulation (taVNS); Device: Physical therapy using Hocoma; Behavioral: Standard of Care

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation (taVNS) — A non-invasive nerve stimulator that stimulates the vagus nerve through the ear.
Device: Physical therapy using Hocoma — Progressive verticalization and mobilization using a robotic tilt table with robotic stepping (Erigo, Hocoma)
Behavioral: Standard of Care — Standard of care with no study interventions. This will include observation of whatever rehabilitation or medical care the patient is currently receiving.

SUMMARY:
Prolonged disorders of consciousness (pDOC) are defined as DOC lasting >1 year post injury for patients with Traumatic Brain Injury (TBI) and >3 months post injury for patients with non-TBI and at present there are limited treatments that reliably lead to enhanced prognosis. The rehabilitation process throughout the continuum of care for patients with pDOC necessitates restorative strategies to facilitate arousal and functional recovery and coordinated medical management. Rehabilitation interventions for patients with DOC and pDOC have evolved in the past decade, with an emerging body of evidence highlighting the benefits of rehabilitation intervention even in the acute. While there is data to support the individual utility of these modalities, no work to date has investigated the benefits of pairing transauricular vagus nerve stimulation (taVNS) and robotic tilt table mobilization (RTTM) to maximize functional recovery in patients with pDOC. This study will report on the safety, feasibility, and preliminary short- and long-term outcomes of RTTM with simultaneously paired Transcutaneous auricular vagus nerve stimulation (taVNS) for Severe Acquired Brain Injury (SABI) patients with pDOC . Fifteen (15) participants will be recruited and complete a 12-week rehabilitation protocol using paired taVNS and RTTM. Once participants have been screened and enrolled in the study, they will complete three study phases: T1: a baseline observation of standard of care T2, intervention, and T3 longitudinal follow up.

DETAILED DESCRIPTION:
T1: At baseline prior to initiating Phase 1, participants will be assessed using Coma Recovery Scale-Revised (CRS-R), Glasgow Coma Scale (GCS), and Glasgow Outcomes Scale- Extended (GOSE). Following this baseline assessment, participants will continue with 4 weeks of their current standard of care. During Phase 1, no study interventions will be implemented. At completion of T1, the CRS-R, GCS, and GOSE will be reassessed. Following Phase 1,

T2a: will be initiated immediately thereby and will entail a 4-week mobilization only phase. Participants will complete 8 sessions of physical therapy over 4 weeks, receiving progressive verticalization and mobilization using a robotic tilt table with robotic stepping (Erigo; Hocoma).

T2b: Immediately after 4 week mobilization only period, participants will complete 8 sessions of physical therapy over 4 weeks, receiving the paired taVNS + RTTM intervention. Upon completion of phase 2b, participants will be reassessed with CRS-R, GCS, and GOSE.

T3: Following the intervention period, participants will complete three additional study visits for assessment at 3-, 6-, and 12-months post intervention using the CRS-R, GOSE, and GCS. Across all study phases, secondary healthcare utilization, including re-admission rates, number of physicians follow up visits and emergency room visits, will be captured from the patient electronic medical record (EMR) and reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of pDOC (includes coma, VS/UWS, MCS, MCS +, MCS-) as defined as disorder of consciousness (DOC) greater than 3 months post onset
* Patients deemed medically safe to participate in physical therapy (PT) as evaluated by the study physicians.

Exclusion Criteria:

* Patients who have emerged from MCS (CRS-R score 6 on Motor Function scale and/or 2 on Communication Scale).
* Patients medically unsafe for participation in PT as indicated by one of the study physicians (including but not limited to those receiving intravenous sedation, those with integumentary breakdown or known pressure injuries, those with cardiovascular or cerebrovascular conditions precluding initiation of physical therapy [ie uncontrolled intracranial pressure, severe symptomatic orthostatic hypotension, etc.).
* Patients with DOC less than 3 months post onset will also be excluded.
* Patients who do not meet technical requirements of the RTTM device will be excluded

  * weighing greater than 135 kg
  * length of legs below 75 cm or above 100 cm,
  * fixed contractures of lower extremity including hip, knee, ankle, or foot).
* Does not have an identified care partner or legally authorized representative to consent to participation

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised (CRS-R) | Baseline, 4 weeks (T1), 8 weeks (T2), and 3-,6-,12-months post intervention (T3)
  The CRS-R is a standardized neurobehavioral rating scale used to monitor recovery of consciousness in persons with severe traumatic brain injury. Six subscales on the CRS-R are summed to provide the total score: auditory function (0-4), visual function (0-5), motor function (0-6), promotor/verbal function (0-3), communication (0-2) and arousal (0-3). Total scores on the CRS-R range from 0 to 23 with high scores generally indicating greater recovery
Glasgow Coma Scale (GCS) | Baseline, 4 weeks (T1), 8 weeks (T2), and 3-,6-,12-months post intervention (T3)
  The Glasgow Coma Scale (GCS) is a reliable and objective way of recording the initial and subsequent level of consciousness in a person after a brain injury. The range of total GCS score is 3 to15 where a higher GCS score represents a better outcome. The scores of subscales are summed to determine the total score*. A GCS score of 13-15 is considered Mild impairment of consciousness; a GCS score of 9-12 is considered Moderate impairment of consciousness; and a GCS score of 3-8 is considered Severe.
  *Subscales:
  * Eyes Response: Spontaneous=4; To sound=3; To Pressure=2; None=1; Not tested
  * Verbal Response: Oriented=5; Confused=4; Words=3; Sounds=2; None=1; Not tested
  * Motor Response: Obeys Commands=6; Localizes=5; Normal Flexion=4; Abnormal Flexion=3; Extension=2; None=1; Not tested
Glasgow Outcomes Scale- Extended (GOSE) | Baseline, 4 weeks (T1), 8 weeks (T2), and 3-,6-,12-months post intervention (T3)
  The GOSE is a scale for functional outcome following a severe traumatic injury. The GOSE is an ordinal variable with the following categories: Dead, Vegetative State, Lower Severe Disability, Upper Severe Disability, Lower Moderate Disability, Upper Moderate Disability, Lower Good Recovery, and Upper Good Recovery. The GOSE score is determined by a structured interview with questions surrounding consciousness, independence inside and outside the home, social and leisure activities and return to normal life among others. The scale is 1-8, level 1 minimum score, level 8 maximum score. A higher score is considered to be a better result. A lower score indicates a worse result.

SECONDARY OUTCOMES:
Readmission Rates | Baseline, 4 weeks (T1), 8 weeks (T2), and 3-,6-,12-months post intervention (T3)
  Readmission Rates
Nociceptive Coma Scale- Revised (NCS-R) | Baseline, 4 weeks (T1), 8 weeks (T2), and 3-,6-,12-months post intervention (T3)
  The NCS-R evaluates behavioral responses to painful stimuli through three subscales: motor, verbal, and facial responses. Each subscale is scored from 0 (no response) to 3 (highest response level), with a total score ranging from 0 to 9, where higher scores indicate greater pain awareness.
Number of Physicians Follow-Up Visits | Baseline, 4 weeks (T1), 8 weeks (T2), and 3-,6-,12-months post intervention (T3)
  Number of Physicians Follow-Up Visits
Number of Emergency Room Visits | Baseline, 4 weeks (T1), 8 weeks (T2), and 3-,6-,12-months post intervention (T3)
  Number of Emergency Room Visits

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Tosto-Mancuso, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Abilities Research Center, Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose.
  Proposals should be directed to AbilitiesResearchCenter@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (to be determined).